CLINICAL TRIAL: NCT00838591
Title: MN-221-CL-007: A Phase II, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of MN-221 When Administered Intravenously as an Adjunct to Standard Therapy to Adults With an Acute Exacerbation of Asthma
Brief Title: Study Evaluating the Safety and Efficacy of MN-221 as an Adjunct to Standard Therapy in Subjects Experiencing an Acute Exacerbation of Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: MediciNova (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MN-221-CL-007
Record Dates: First submitted 2009-02-05; First posted 2009-02-06 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Asthma
Keywords: MN-221; Asthma; Acute; Exacerbation
MeSH Terms: conditions — Asthma | interventions — bedoradrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): MN-221 given i.v. 1-hour infusion a total dose of 1200 μg (40 μg/min for 15 min [600 μg] + 13.3 μg/min for 45 min [600 μg]) as an adjunct to the standard of care for acute exacerbation of asthma.
  Interventions: Drug: MN-221
- Placebo (Placebo Comparator): Placebo (Lot #CLO-095) was packaged in identical vials containing only excipients and administered as an i.v. 1-hour infusion with a regimen as described for MN-221.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MN-221 — Dose: intravenous 1-hour infusion of MN-221 (total dose 1200 μg) or matching placebo.
  Other Names: bedoradrine sulfate
  Arms: 1
Drug: Placebo
  Arms: Placebo

SUMMARY:
The objective of this clinical study is to examine the safety and effectiveness of intravenous MN-221 compared to placebo when administered as an adjunct to standard therapy in subjects experiencing an acute exacerbation of asthma.

DETAILED DESCRIPTION:
This is an international, randomized, double-blind, placebo-controlled, multi-center ED study. Each subject will receive MN-221 or placebo administered through a continuous intravenous infusion in addition to the standardized treatment for an acute exacerbation of asthma.

Upon presentation to the ED for assessment and treatment for an acute exacerbation of asthma the patient should receive standard of care consistent with the international guidelines (e.g., Global Initiative for Asthma [GINA] or the National Asthma Education and Prevention Program [NAEPP]) and required, in part, by this protocol prior to screening procedures being performed.

Prior to any study specific treatment or evaluation being performed a subject must have signed an IRB/EC/REB approved consent form. Once the subject has received the initial treatment regimen the subject will be assessed for response to the treatment including spirometry.If the subject meets all entry criteria the subject will be randomized to receive MN-221 or placebo. Throughout the screening process the subject will continue to receive standardized treatment consistent with the appropriate guidelines for the treatment of acute exacerbations of asthma.

Subjects enrolled in the study will receive an intravenous 1-hour infusion of MN-221 study drug or placebo. Subjects receiving MN-221 will be administered a total dose of 1200 μg.

During the study treatment period, the subject may continue to receive standardized treatment and be assessed. The study treatment period will be approximately 3 hours in length. Safety and efficacy will be monitored throughout the treatment period. PK parameters (if applicable) will be obtained from subjects at selected study sites. A blood sample for genomic evaluation will be collected during the treatment period (at participating sites) if the subject consents to the evaluation. An initial 24-hour post-randomization follow-up visit will be completed to evaluate the subject's health status as well as for safety and PK parameters (if applicable). A second follow-up contact will be completed by telephone seven days post-randomization for safety purposes and to evaluate the subject's health status.

A periodic risk/benefit evaluation will be performed by the study's Data Safety Monitoring Board.

ELIGIBILITY:
Inclusion Criteria:

* Subjects meeting all of the following criteria will be considered for admission to the study:

  1. Male or female 18 to 65 years of age, inclusive;
  2. Self-reported history of physician-diagnosed and treated asthma for ≥ 3 months prior to randomization;
  3. A diagnosis of an acute exacerbation of asthma upon presentation at the ED as defined by dyspnea and evidence of bronchospasm;
  4. Received the following Standardized Treatment within a 2-hour time window and prior to obtaining the Qualifying Spirometry value(FEV1):

     * Supplemental oxygen given to maintain oxygen saturation as measured by pulse oximetry of ≥ 90% as needed;
     * Albuterol 5-15mg of albuterol via nebulizer prior to the qualifying spirometry evaluation; simultaneously with
     * Ipratropium 0.5-1.5 mg of ipratropium via nebulizer prior to the qualifying spirometry evaluation;
     * One dose of corticosteroid of at least 50 mg given orally (prednisone) or intravenously (methylprednisolone) or the equivalent dose of another corticosteroid.
  5. FEV1 of ≤ 50% of predicted; NOTE: Spirometry to measure the subject's FEV1 expressed as % of predicted within 30 minutes of completing administration of 5 mg (but not more than 15 mg) albuterol and 0.5 mg (but not more than 1.5 mg) of ipratropium..
  6. Negative urine pregnancy test for all females of child-bearing potential;
  7. ECG with no dysrhythmias (except sinus tachycardia);
  8. No clinical or electrocardiographic signs of ischemic heart disease as determined by the Investigator; and
  9. Legally effective written informed consent obtained prior to starting any mandated study procedures

Exclusion Criteria:

Subjects will be excluded if they meet any of the following criteria:

1. Administration of a parenteral (intravenous or subcutaneous) beta agonist (e. g., albuterol, terbutaline, epinephrine) within 6 hours prior to randomization;
2. A current or prior diagnosis or suspected diagnosis of COPD or other chronic lung disease other than asthma;
3. Presence of pneumonia;
4. Presence of significant other respiratory dysfunction such as pneumothorax, pneumomediastinum, or pulmonary edema;
5. Known or suspected vocal cord dysfunction syndrome;
6. Presence of aspirated foreign body (known or suspected);
7. History or any current clinical evidence suggesting cardiomyopathy or congestive heart failure;
8. History or presence of tachyarrhythmias, with the exception of sinus tachycardia;
9. Heart rate ≥ 140 bpm;
10. Hypokalemia, defined as subjects with serum potassium level of <2.8 mEq/L (≤2.8 mmol/L) obtained at Screening (local stat lab, blood gas analysis, or other point of care device) with the following exception:

    For the subjects using non-potassium-sparing diuretics (i.e. loop-diuretic or thiazide diuretic) without "potassium-sparing diuretics" (e.g., Triamterene or Spironolactone) OR without potassium supplementation of at least KCl 20 mEq/day whose potassium level <3.5 mEq/L (<3.5 mmol/L) at Screening.
11. Significant cardiac, renal, hepatic, endocrine, metabolic, neurologic or other systemic disease. A significant disease will be defined as one which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study or the subject's ability to participate in the trial;
12. Self-reported history of greater than 20 pack-yr smoking history;
13. Fever ≥ 102.0 ºF (38.9 ºC);
14. Uncontrolled hypertension defined as a blood pressure ≥ 170/100 mm Hg (22.7/13.3 kPa);
15. Need for immediate intubation, mechanical ventilation, or non-invasive positive pressure ventilation as determined by the Investigator;
16. Pregnant or lactating females;
17. Participated in another clinical study with an investigational drug within 30 days of randomization;
18. Positive urine drug screen for cocaine, methamphetamine or PCP unless, in the Investigator's clinical judgment, a single positive result is explained by exposure to a non-illicit drug product (i.e., is a false positive). For example, phenylpropanolamine or methylphenidate may read positive in a methamphetamine screen; dextromethorphan in a PCP screen.
19. Any subject with a known allergy to components of the MN-221 drug product;
20. Any subject with a known allergy to other beta agonists;
21. Previous exposure to MN-221; or
22. Use of theophylline, beta blockers, digoxin, MAO inhibitors, or tricyclic antidepressants within 2 weeks prior to randomization.

Use of non-potassium-sparing diuretics (i.e. Thiazide or Loop-diuretic) without potassium-sparing diuretic OR without potassium supplementation >20 mEq/day within 2 weeks prior to randomization and if serum potassium level at Screening <3.5 mEq/L (<3.5 mmol/L).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2009-03; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
The primary efficacy analysis will be based on a change in FEV1, expressed as percent of predicted, at Hour 3 when compared to FEV1, expressed as percent of predicted, at the qualifying/screening timepoint. | Hour 3

SECONDARY OUTCOMES:
Change from baseline FEV1 % of predicted (at time points other than Hour 3) | Hours 1, 2, 3, and 24
Change from baseline FEV1 (L) | Hours 1, 2, 3 and 24
Change from baseline PEFR (L/sec) | Hours 1, 2, 3 and 24
Change from baseline PEFR, expressed as percent (%) of predicted | Hours 1, 2, 3and 24
Improvement in Dyspnea index scale | Hours 1, 2, 3, 24 and Day 8
Percent of subjects with an improvement in FEV1 ≥ 200cc | Hours 1, 2, 3 and 24
Percent of subjects with an improvement in FEV1, % predicted ≥ 5% | Hours 1, 2, 3 and 24
Percent of subjects with and improvement in FEV1, % predicted ≥ 10% | Hours 1, 2, 3 and 24
Subjects Hospitalized ( within 24 hour from start of study drug infusion) | Within 24 hours from start of study drug infusion.
Admitted to ICU (within 24 hours from start of study drug infusion) | Within 24 hours from start of study drug infusion.
Number of albuterol treatments to achieve an increase in FEV1% of predicted ≥ 15% | Hours 3
Total dose or number of albuterol treatments in first 3 hours following commencement of randomized medication. | No specific time points
Time to achieve an increase of FEV1% of predicted ≥ 15% | No specific time points
Time to initial albuterol treatment following the commencement of randomized medication | No specific time points
Hospital length of stay | No specific timepoints

CONTACTS AND LOCATIONS:
Overall Officials: Kazuko Matsuda, MD, Study Director — MediciNova
Locations (15):
- United States (15):
  - Loma Linda University Medical Center, Loma Linda, California
  - UCSD Medical Center - Thornton Hospital, San Diego, California
  - UCSD Medical Center, San Diego, California
  - Olive View - UCLA Medical Center, Sylmar, California
  - Loyola University Medical Center, Maywood, Illinois
  - Newton - Wellesley Hospital, Newton, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - University of Cincinnati, Cincinnati, Ohio
  - Albert Einstein Healthcare Network, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Sentara General Hospital, Norfolk, Virginia

REFERENCES:
- [Derived] House SL, Matsuda K, O'Brien G, Makhay M, Iwaki Y, Ferguson I, Lovato LM, Lewis LM. Efficacy of a new intravenous beta2-adrenergic agonist (bedoradrine, MN-221) for patients with an acute exacerbation of asthma. Respir Med. 2015 Oct;109(10):1268-73. doi: 10.1016/j.rmed.2015.08.003. Epub 2015 Aug 14. PMID 26324315
- [Derived] Schneider JE, Lewis LM, Ferguson I, House SL, Liu J, Matsuda K, Johnson K. Repeated dyspnea score and percent FEV1 are modest predictors of hospitalization/relapse in patients with acute asthma exacerbation. Respir Med. 2014 Sep;108(9):1284-91. doi: 10.1016/j.rmed.2014.06.006. Epub 2014 Jul 8. PMID 25087835